CLINICAL TRIAL: NCT01800773
Title: Written Exposure Therapy for Post Traumatic Stress Disorder: A Randomized Noninferiority Trial
Brief Title: Written Exposure Therapy for Posttraumatic Stress Disorder
Acronym: WET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-31806; 1R01MH095737-01A1 (NIH)
Record Dates: First submitted 2013-02-15; First posted 2013-02-28 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; exposure treatment; clinical trial; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Exposure Therapy (Experimental): Written exposure treatment is a 5 session treatment in which participants write about their trauma event in a specified manner.
  Interventions: Behavioral: Written Exposure Therapy
- Cognitive Processing Therapy (Active Comparator): cognitive processing therapy will be included as the evidence-based treatment for PTSD in this study.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Written exposure therapy is a 5 session, weekly treatment in which individuals write about their trauma event in a specified manner.
  Arms: Written Exposure Therapy
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy (CPT) is an evidence-based treatment for PTSD. CPT consists of 12, weekly sessions.
  Arms: Cognitive Processing Therapy

SUMMARY:
Although evidence-based treatments for PTSD exist, a significant minority of individuals do not benefit from these treatments and many individuals to not seek treatment, citing barriers such as time commitment and expense of treatment. The goal of the proposed study is to establish an alternative PTSD treatment that is efficacious and efficient.

DETAILED DESCRIPTION:
Prior research has demonstrated that written exposure therapy (WET), is an efficient, well-tolerated, and efficacious treatment for PTSD. The proposed project takes the next step in establishing WET as an intervention for PTSD by examining whether WET is equally efficacious to an evidence-based treatment for PTSD. Using a randomized noninferiority controlled trial, 126 adults diagnosed with PTSD will be assigned to either WET or Cognitive Processing Therapy (CPT). Outcome data will be collected at baseline and 6-, 12-, 24-, 36- and 60-weeks post-first treatment session. The primary aim is to examine whether PTSD participants assigned to WET demonstrate PTSD symptom severity outcome that is noninferior to PTSD participants assigned to CPT. Secondary aims include examining whether expected treatment gains are sustained for both treatments and whether WET has a lower treatment dropout rate relative to CPT. Exploratory aims include examining moderators and mediators of WET and CPT. If the hypothesis that WET is noninferior to CPT is confirmed then a brief treatment option for PTSD will be established.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis
* if taking psychotropic medication, on stable dose for 2 months
* Ability to read and write in English

Exclusion Criteria:

* not currently engaged in active PTSD treatment
* no current diagnosis of substance dependence
* no current diagnosis of psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-03-09 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | change from baseline PTSD symptom severity at 36 weeks post first treatment session
  Total score on the CAPS will be used to assess change in PTSD symptom severity from baseline (pre-treatment) until 36- weeks post first treatment session.

SECONDARY OUTCOMES:
treatment dropout | course of treatment
  Treatment condition differences in treatment drop out rate at post-treatment (treatment duration is 5 weeks for WET condition and 12 weeks for CPT condition).

CONTACTS AND LOCATIONS:
Overall Officials: Denise M. Sloan, Ph.D., Principal Investigator — Boston University
Locations (1):
- National Center for PTSD at VA Boston Healthcare System, Boston, Massachusetts, United States

REFERENCES:
- [Result] Sloan DM, Marx BP, Lee DJ, Resick PA. A Brief Exposure-Based Treatment vs Cognitive Processing Therapy for Posttraumatic Stress Disorder: A Randomized Noninferiority Clinical Trial. JAMA Psychiatry. 2018 Mar 1;75(3):233-239. doi: 10.1001/jamapsychiatry.2017.4249. PMID 29344631